CLINICAL TRIAL: NCT05515809
Title: Evaluation of the Effect of Para-sternal Block on Postoperative Respiratory Function After Cardiac Sternotomy Surgery
Acronym: PARACARD
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI2021_843_0229
Record Dates: First submitted 2022-07-28; First posted 2022-08-25 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Cardiac Surgery; Ultrasound-guided Parasternal Block; Postoperative Pulmonary Complications; Pulmonary Function Testing
Keywords: Cardiac surgery; Ultrasound-guided Parasternal Block; Postoperative pulmonary complications; Pulmonary function testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- interventional arm (Experimental): the experimental arm will receive the parasternal block with injection of locoregional anesthesia
  Interventions: Drug: parasternal block
- control arm not requiring loco-regional anesthesia. (Active Comparator): the control arm will receive a standard treatment, without locoregional anesthesia
  Interventions: Drug: Standard pain management

INTERVENTIONS:
Drug: parasternal block — Echo-guided loco-regional anesthesia by bilateral parasternal block in immediate preoperative.
  The drug used is Ropivacaine 2mg/ml, 0.2%. Injection of 20ml per side, under ultrasound control, after general anaesthesia and before skin incision, and therefore before surgery
  Arms: interventional arm
Drug: Standard pain management — Standard pain management care involves a multimodal strategy that includes the use of intravenous analgesics. Morphine medications are the mainstay of pain management
  Arms: control arm not requiring loco-regional anesthesia.

SUMMARY:
Postoperative pain after cardiac surgery is associated with reduced postoperative respiratory function. There is an association between greater pain and more pronounced decreases in lung volumes postoperatively. With an incidence of 10% to 25% of cases, pulmonary complications are the second source of postoperative morbidity after cardiac complications; in 2-5% of cases, the dysfunction is severe and leads to significant consequences that can lead to death. It has been shown that postoperative pain after cardiac surgery is associated with a reduction in functional respiratory capacity. There is an association between greater pain and more pronounced decreases in lung volumes postoperatively. The main objective of this study will be to evaluate the impact of locoregional anesthesia by parasternal block analgesic on postoperative respiratory function at D1 postoperatively

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Elective cardiac surgery under CEC with sternotomy
* Written informed consent from the patient.
* Women of childbearing age must have a negative urine HCG pregnancy test.

Exclusion Criteria:

* Thoracotomy approach
* Mini-sternotomy approach
* Opioid drug dependence or chronic opioid drug use
* Chronic benzodiazepine use (respiratory depressant treatment or treatment that may affect postoperative respiratory function)
* Contraindication or allergy to local anesthetics
* Emergency surgery
* Acute infective endocarditis
* Immunosuppressive or steroid treatment (prednisone > 0.5mg/kg/day or equivalent)
* AIDS with CD4 count <200/mm3
* Autoimmune disorder
* Transplant recipient
* Inclusion in another study within the last 30 days.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-07-19 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Change in postoperative forced vital capacity (FVC) | 1 day
  The primary endpoint was the change (reduction) in postoperative forced vital capacity (FVC) between the preoperative measurement and at D1 postoperatively.
  * "Forced Vital Capacity measured by SPIROLAB spirometry (Appendix).
  * "Vital capacity is expressed as % of theoretical value.

SECONDARY OUTCOMES:
Variation of FCV between both groups | at day 2
  Respiratory functional investigations at day 2 is forced vital capacity (FVC)
Variation of FCV between both groups | at 1 month
  Respiratory functional investigations at 1 month is forced vital capacity (FVC)
Variation of FCV between both groups | at 3 months
  Respiratory functional investigations at 3 months is forced vital capacity (FVC)
Variation of forced expiratory volume in 1 second (FEV1) | at day 2
  Respiratory functional investigations at day 2 are forced expiratory volume in 1 second (FEV1)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens-Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: No